CLINICAL TRIAL: NCT05301790
Title: Added Value of Breast MRI in Evaluation of Pathologic Response in Patients With Locally Advanced Breast Cancer Who Undergo Neoadjuvent Chemotherapy
Brief Title: Breast MRI in Evaluation of Pathologic Response in Patients With Breast Cancer With Neoadjuvent Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Maher Ebied Maher, resident, Assiut University
Other Study IDs: MRI in breast cancer
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Role of MRI in Evaluation of Breast Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — use of MRI modality of imaging in evaluation of pathologic response in patients with breast cancer

SUMMARY:
evaluation of pathological response in breast mass by use of breast MRI in patients receiving neoadjuvent chemotherapy via comparison with pathological results

DETAILED DESCRIPTION:
evaluation of pathological response in locally advanced breast masses by use of breast MRI in patients receiving neoadjuvent chemotherapy via comparison with pathological results

ELIGIBILITY:
Inclusion Criteria:

* all women referred to the radiology department for breast MRI examination either for screening, evaluation of suspicious lesions onsono-mammography \

  * Patients with locally advanced breast cancer
  * Patients with early stage breast cancer and chemo-responsive tumour markers (i.e. triple negative, Her2+), who will benefit from downsizing for breast conserving surgery (BCS)
  * Absolute or Relative contraindications to surgery (advanced age/multiple medical comorbidities) in the setting of estrogen receptor positive tumours (for consideration of neoadjuvant endocrine therapy)3
  * Patients must be elder than 18 years old.
* patients with accepted renal function

Exclusion Criteria:

* Patients with metastatic breast cancer.
* Patient with breast mass more than 5 cm .
* Patients with fungating breast mass .
* Patients with stage IV [tumor spread to chest wall and to skin ].
* pregnant women especially in 1th trimester.
* Patient with presence of any paramagnetic substance as pacemakers.
* severely ill patients .
* patients with claustrophobia.
* arrhythmic patients

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: * all women referred to the radiology department for breast MRI examination either for screening, evaluation of suspicious lesions onsono-mammography \
    * Patients with locally advanced breast cancer
    * Patients with early stage breast cancer and chemo-responsive tumour markers (i.e. triple negative, Her2+), who will benefit from downsizing for breast conserving surgery (BCS)
    * Absolute or Relative contraindications to surgery (advanced age/multiple medical comorbidities) in the setting of estrogen receptor positive tumours (for consideration of neoadjuvant endocrine therapy)3
    * Patients must be elder than 18 years old.
  * patients with accepted renal function
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
comparison of MRI findings with pathologic results | baseline
  added value of breast MRI in evaluation of pathologic response in patients with locally advanced breast cancer who undergo neoadjvent chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: lamiaa mohamed refaat, assisstant professor, Study Director — assiut university -south egypt cancer institute; omar mostafa, lecturer, Study Director — assiut university-south egypt cancer institute

IPD SHARING:
Plan to Share IPD: No